CLINICAL TRIAL: NCT01384227
Title: Evaluation of a Miniaturized Microscope Device for the Detection of Barrett's Neoplasia: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anandasabapathy, Sharmila, M.D. (Individual)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Sharmila Anandasabapathy, MD, Associate Professor of Medicne, Anandasabapathy, Sharmila, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: GCO # 08-1190; NCT00755625 (obsolete NCT alias)
Record Dates: First submitted 2011-06-21; First posted 2011-06-29 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's esophagus; in vivo imaging; image guide microscope
MeSH Terms: conditions — Barrett Esophagus | interventions — Proflavine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proflavine Hemisulfate (Experimental)
  Interventions: Drug: Proflavine Hemisulfate

INTERVENTIONS:
Drug: Proflavine Hemisulfate — Proflavine hemisulfate 0.01% (derived from dissolving 10 mg Proflavine Hemisulfate USP in 100 ml of sterile water)
  Other Names: Proflavine

SUMMARY:
The overall objective of this study is to obtain data to evaluate whether high-resolution imaging of barrett's esophagus in vivo can assist clinicians in detecting dysplastic (precancerous) areas. This is a pilot study of an novel technology, a miniaturized microscope device which can be used during upper endoscopy to image the gastrointestinal epithelium. This is an exploratory, not a comparative, study designed to evaluate the feasibility of using this instrument in Barrett's esophagus.

ELIGIBILITY:
Inclusion Criteria:

* Barrett's without dysplasia
* Barrett's with dysplasia
* Esophageal Adenocarcinoma

Exclusion Criteria:

* Subjects unfit for standard upper endoscopy
* Subjects currently receiving chemo or radiation treatment
* Subject currently receiving PDT or ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-02; Primary Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To determine whether tissue is neoplastic or non-neoplastic | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Anandasabapathy, Principal Investigator — Mt. Sinai School of Medicine
Locations (1):
- Mount Sinai Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Shin D, Lee MH, Polydorides AD, Pierce MC, Vila PM, Parikh ND, Rosen DG, Anandasabapathy S, Richards-Kortum RR. Quantitative analysis of high-resolution microendoscopic images for diagnosis of neoplasia in patients with Barrett's esophagus. Gastrointest Endosc. 2016 Jan;83(1):107-14. doi: 10.1016/j.gie.2015.06.045. Epub 2015 Aug 5. PMID 26253018